CLINICAL TRIAL: NCT03166722
Title: Cerebral Regional Tissue Oxygen Saturation to Guide Oxygen Delivery in Preterm Neonates During Immediate Transition After Birth: An Investigator-initiated Randomised Multi-centre Multinational Clinical Trial
Brief Title: Cerebral Regional Tissue Oxygen Saturation to Guide Oxygen Delivery in Preterm Neonates During Immediate Transition
Acronym: COSGOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Royal Alexandra Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: COSGOD Phase III
Record Dates: First submitted 2017-05-03; First posted 2017-05-25 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Preterm Infant; Brain Injuries; Birth Hypoxia
MeSH Terms: conditions — Premature Birth; Brain Injuries | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: investigator-initiated randomised multi-centre multinational clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group: Invos 5100 (Experimental): Supplemental oxygen support and respiratory/circulatory support is guided by cerebral regional tissue oxygenation (crSO2) measured with near-infrared spectroscopy ("INVOS 5100" ), in addition to the SpO2/HR (oxygen saturation/heart rate) monitoring according to routine.
  Interventions: Device: Study group
- Control group: Routine care (Active Comparator): Supplemental oxygen support and respiratory/circulatory support is guided by SpO2/HR monitoring according to routine - The resuscitation team is blinded to the crSO2 monitoring.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Control group — SpO2 and HR monitoring and routine treatment during immediate transition
  Arms: Control group: Routine care
Device: Study group — Cerebral NIRS measurement with INVOS 5100 during immediate transition in addition to SpO2 and HR monitoring
  Arms: Study group: Invos 5100

SUMMARY:
The aim of the COSGOD Phase III trial is to examine, if it is possible to increase survival without cerebral injury in preterm neonates <32 weeks of gestation by monitoring the cerebral tissue oxygen saturation in addition to routine monitoring of arterial oxygen saturation and heart rate and specified clinical treatment guidelines during immediate transition period after birth (the first 15 minutes).

DETAILED DESCRIPTION:
Background

The transition to life after birth is a complex physiological process where the neonate has to establish sufficient ventilation and changes from intra-uterine circulation to extra-uterine circulation take place. During these processes the neonate has to provide the brain with adequate perfusion and oxygen delivery to maintain normal cerebral tissue oxygenation and activity. If hypoxia and bradycardia both common events during immediate transition in preterm neonates occur, cerebral hypoxia-ischaemia may cause perinatal brain injury that is the major causes of mortality and long term neurodevelopmental impairment.

Objectives

The primary objective of the COSGOD Phase III trial is to examine, if it is possible to increase survival without cerebral injury in preterm neonates <32 weeks of gestation by monitoring the cerebral tissue oxygen saturation in addition to routine monitoring of arterial oxygen saturation (SpO2) and heart rate (HR) and specified clinical treatment guidelines during immediate transition period after birth (the first 15 minutes).

Hypothesis

The investigators hypothesise that using cerebral tissue oxygen saturation in addition to SpO2 and HR monitoring and specified treatment guidelines during immediate transition and resuscitation would increase survival without cerebral injury in preterm neonates.

Trial design

An investigator-initiated randomised, multi-centre, multinational, phase III clinical trial involving preterm infants from European countries and North America.

Inclusion and exclusion criteria

The inclusion criteria are: neonates born more than 8 weeks preterm (gestational age up to 31 weeks and 6 days); decision to conduct full life support; parental informed consent; and cerebral NIRS oximeter placed within three minutes after birth.

Sample size

According to actual data of two European centres (Graz and Rotterdam) and one Canadian centre (Edmonton) the percentage of neonates not affected by mortality and cerebral injury is 65%. Assuming an increase of not affected neonates from 65% to 75% and a dropout rate of 10% a total of 724 neonates are required to detect this difference with a two group χ² test (alpha: 0.05, power: 80%).

Intervention

The premature infants will be randomised into experimental or control group. Both groups will have a near infrared spectroscopy (NIRS) device (left frontal), pulse-oximeter (right wrist) and electrocardiogram placed within three minutes after birth. In the study group, the cerebral tissue saturation, SpO2 and HR readings are visible, and the infant will be treated accordingly using a defined treatment guideline. In the control group, only SpO2 and HR will be visible, and the infant will be treated according routine treatment.

Duration of intervention Monitoring will be started within 3 minutes after birth and the intervention will last during immediate transition period and resuscitation up to 15 minutes after birth.

Follow up

Thereafter, each neonate will be followed up for primary outcome to term date or discharge.

Outcome measures

The primary outcome is mortality and/or cerebral injury defined as any intraventricular bleeding and/or cystic periventricular leucomalacia.

The secondary outcomes are neonatal morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates less than completed 32 weeks,
* Decision to conduct full life support,
* Written informed consent.

Exclusion Criteria:

* No decision to conduct full life support,
* No written informed consent,
* Congenital malformation.

Ages: 1 Minute to 15 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 655 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Mortality and/or occurrence of cerebral injury | up to 19 weeks after birth
  Number of patients, who die or have intraventricular hemorrhage or have periventricular leucomalacia

SECONDARY OUTCOMES:
Frequency of neonatal morbidities | up to 19 weeks after birth
  Number of patients, who have infection and/or sepsis and/or necrotizing enterocolitis bronchoplumonary dysplasia, retinopathia prematurorumand/or bronchoplumonary dysplasia and /or retinopathia prematurorum
Sex | up to 19 weeks after birth
  Number of male and female patients, who die or have intraventricular hemorrhage or have periventricular leucomalacia
Gestational age | up to 19 weeks after birth
  Number of patients with less than 28 weeks of gestation and more than or equal 28 weeks of gestation, who die or have intraventricular hemorrhage or have periventricular leucomalacia

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Pichler, MD, Principal Investigator — Medical University of Graz, Austria; Georg M Schmölzer, MD, PhD, Principal Investigator — Royal Alexandra Hospital, Edmonton, Canada
Locations (12):
- Austria (3):
  - Department of Pediatrics, Medical University of Graz, Graz, Styria
  - Medical University Innsbruck, Innsbruck
  - Medical University Vienna, Vienna
- Royal Alexandra Hospital, Edmonton, Alberta, Canada
- Germany (2):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Centre for Pediatric Clinical Studies, Tübingen
- University College Cork, Cork, Ireland
- Italy (2):
  - Ospedale dei Bambini "V.Buzzi" Milano, Milan
  - Institute for Maternal and Child Health, IRCCS Burlo Garofolo, Trieste
- Poland (2):
  - Poznan University of Medical Sciences, Poznan
  - Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
The demographic data and data of primary and secondary outcome will be stored at and available form the Institut for Medical Informatics, Statistics und Documentation, Medical University of Graz, Austria
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of primary and secondary outcome
Access Criteria: On demand

REFERENCES:
- [Derived] Perme T, Kornhauser Cerar L, Schwaberger B, Urlesberger B, Wolfsberger CH, Baik N, Goeral K, Hammerl M, Dempsey EM, Springer L, Lista G, Szczapa T, Fuchs H, Karpinski L, Bua J, Avian A, Law BHY, Buchmayer J, Kiechl-Kohlendorfer U, Schwarz CE, Gruendler K, Stucchi I, Klebermass-Schrehof K, Schmolzer GM, Pichler G; COSGOD III study group. Effect of timing of umbilical cord clamping on cerebral regional tissue oxygenation: a secondary analysis of the COSGOD III trial. Arch Dis Child Fetal Neonatal Ed. 2025 Oct 17;110(6):610-615. doi: 10.1136/archdischild-2024-327946. PMID 40306760
- [Derived] Pichler G, Goeral K, Hammerl M, Perme T, Dempsey EM, Springer L, Lista G, Szczapa T, Fuchs H, Karpinski L, Bua J, Avian A, Law B, Urlesberger B, Buchmayer J, Kiechl-Kohlendorfer U, Kornhauser-Cerar L, Schwarz CE, Grundler K, Stucchi I, Schwaberger B, Klebermass-Schrehof K, Schmolzer GM; COSGOD III study group. Cerebral regional tissue Oxygen Saturation to Guide Oxygen Delivery in preterm neonates during immediate transition after birth (COSGOD III): multicentre randomised phase 3 clinical trial. BMJ. 2023 Jan 24;380:e072313. doi: 10.1136/bmj-2022-072313. PMID 36693654
- [Derived] Pichler G, Baumgartner S, Biermayr M, Dempsey E, Fuchs H, Goos TG, Lista G, Lorenz L, Karpinski L, Mitra S, Kornhauser-Cerar L, Avian A, Urlesberger B, Schmolzer GM. Cerebral regional tissue Oxygen Saturation to Guide Oxygen Delivery in preterm neonates during immediate transition after birth (COSGOD III): an investigator-initiated, randomized, multi-center, multi-national, clinical trial on additional cerebral tissue oxygen saturation monitoring combined with defined treatment guidelines versus standard monitoring and treatment as usual in premature infants during immediate transition: study protocol for a randomized controlled trial. Trials. 2019 Mar 20;20(1):178. doi: 10.1186/s13063-019-3258-y. PMID 30894226